CLINICAL TRIAL: NCT07204275
Title: A Phase 2b/3 Adaptive, Randomized, Active-controlled Study Evaluating the Efficacy, Safety, and Tolerability of Povetacicept Versus Calcineurin Inhibitor in the Treatment of Primary Membranous Nephropathy
Brief Title: A Study to Evaluate Efficacy, Safety, and Tolerability of Povetacicept in Participants With Primary Membranous Nephropathy (pMN)
Acronym: OLYMPUS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX24-AIS-D10; 2025-521661-27-00 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 2b: Povetacicept (Experimental): Participants will be randomized to receive one of the two doses of Povetacicept.
  Interventions: Drug: Povetacicept
- Phase 3: Povetacicept (Experimental): Participants will be randomized to receive one of the two doses of Povetacicept (dose selected based on Phase 2b).
  Interventions: Drug: Povetacicept
- Phase 3: Calcineurin Inhibitor (CNI) (Active Comparator): Participants will be randomized to receive the calcineurin inhibitor (CNI) Tacrolimus.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Povetacicept — Solution for Subcutaneous Injection.
  Arms: Phase 2b: Povetacicept; Phase 3: Povetacicept
Drug: Tacrolimus — Capsules for Oral Administration.
  Arms: Phase 3: Calcineurin Inhibitor (CNI)

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of povetacicept in participants with primary membranous nephropathy (pMN).

ELIGIBILITY:
Key Inclusion Criteria:

• Diagnosed with pMN with confirmatory historical biopsy. If no historical biopsy was performed that confirmed pMN, a biopsy can be performed during Screening to confirm eligibility

Key Exclusion Criteria:

• Hypersensitivity to investigational medicinal product or to any of its excipients

Other protocol defined Inclusion/Exclusion criteria will apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-12-29 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Complete Clinical Remission Definition 1 (CR1) | At Week 104

SECONDARY OUTCOMES:
Proportion of Participants with Complete Clinical Remission Definition 2 (CR2) | At Week 104
Proportion of Participants with Overall Clinical Remission (OR) | At Week 104

CONTACTS AND LOCATIONS:
Locations (38):
- United States (22):
  - Renal Associates, Montgomery, Alabama
  - Southwest Kidney Institute, PLC (SKI) - Surprise, Surprise, Arizona
  - Academic Medical Research Institute (AMRI), Los Angeles, California
  - Valiance Clinical Research - Internal Medicine, Tarzana, California
  - Western Nephrology & Metabolic Bone Disease PC, Arvada, Colorado
  - Bioresearch Partner, Miami, Florida
  - CTR Oakwater, LLC, Orlando, Florida
  - Clinical Site Partners, LLC - Orlando, Winter Park, Florida
  - DaVita Clinical Research Columbus, Columbus, Georgia
  - Georgia Nephrology, Lawrenceville, Georgia
  - CARE Institute-Boise Kidney, Boise, Idaho
  - NANI Research, Hinsdale, Illinois
  - DaVita Clinical Research Edina, Edina, Minnesota
  - Kidney Specialists of Southern Nevada, Las Vegas, Nevada
  - Carolina Nephrology Greenville, Greenville, South Carolina
  - Carolina Nephrology, PA, Spartanburg, South Carolina
  - El Paso Kidney Specialists, El Paso, Texas
  - Provecta Research Network, Houston, Texas
  - DaVita Clinical Research Houston, Houston, Texas
  - Davita Clinical Research San Antonio, San Antonio, Texas
  - Utah Kidney Research, Salt Lake City, Utah
  - Milwaukee Neprologists, SC, Wauwatosa, Wisconsin
- China (16):
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Sichuan Academy of Medical Sciences ＆ Sichuan Provincial People's Hospital, Chengdu
  - Dalian Municipal Central Hospital, Dalian
  - Fuyang People's Hospital, Fuyang
  - Guangdong Provincial People's Hospital, Guangzhou
  - The Affiliated Huai'an No.1 People's Hospital of Nanjing Medical University, Huai'an
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Nanyang Central Hospital, Nanyang
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Wuxi People's Hospital, Wuxi
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Yantai YuHuangDing Hospital, Yantai
  - Yichang Central People Hospital, Yichang

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/